CLINICAL TRIAL: NCT06220344
Title: Honey Dressing - A Preventive Procedure for Post-Surgical Site Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Syed Muhammad Ali Haider, House Officer Neurosurgery, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HITEC-IMS-01-2022
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Wound Infection; Wound Dehiscence; Wound Bleeding; Wound Surgical
MeSH Terms: conditions — Wound Infection; Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey (Experimental): Participants will get honey dressings in their follow-up visits to the dressing room.
  Interventions: Biological: Honey Dressing
- Aseptic Iodine (Active Comparator): Participants will get iodine solution dressings in their follow-up visits to the dressing room.
  Interventions: Drug: Iodine Dressing

INTERVENTIONS:
Biological: Honey Dressing — Honey Dressing will be applied from the 1st Post-Op day till the fully healed wound, which is described as no dehiscence, no exudate, no warmth, and sutures removed.
  Arms: Honey
Drug: Iodine Dressing — Iodine Dressing will be applied from the 1st Post-Op day till the fully healed wound, which is described as no dehiscence, no exudate, no warmth, and sutures removed.
  Other Names: Iodine solution dressing
  Arms: Aseptic Iodine

SUMMARY:
The goal of this clinical trial is to compare the wound healing in the participants who underwent the clean surgical procedure, by applying honey dressing and common Iodine solution dressing, participants will have no other co-morbidities like Diabetes, Anemia, etc. which can make the results biased. The main questions it aims to answer are:

* Do the iodine solutions are enough to counter the infections caused by resistant strains of bacteria?
* What is the efficacy and efficiency of honey dressing in wound care?

Participants will be tasked to

* Ensure strict follow-up in the hospital dressing room
* Half of the participants will apply common iodine solution dressing and the other half will be applied honey dressing.

Researchers will compare Iodine dressing (Control group) with Honey dressing (Experimental group) to see if Honey dressing is better in the prevention of post-surgery wound infection and if it is cost-efficient and its efficacy.

ELIGIBILITY:
Inclusion Criteria:

Patients with sterile/clean post-surgical wounds are admitted in general surgery, neurosurgery, orthopedic, and gynecology wards and require follow-up dressings.

Exclusion Criteria:

1. Patients with:

   * Anemia
   * BMI>30
   * Local Infection in wound area.
   * Venous leg ulcers
   * Diabetes
   * Immunocompromised (Oncological patients)
2. Patient under negative pressure therapy

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Signs of Wound Infection | 3rd day, 7th day, 15th day.
  Presence of exudate, warmth, pus, erythema, dehiscence, contact bleeding, and any systemic sign like fever, rash, and myalgia.

CONTACTS AND LOCATIONS:
Locations (1):
- Heavy Industry Taxila Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No